CLINICAL TRIAL: NCT01877239
Title: A Multicenter Non-interventional Study To Observe The Safety And Efficacy Of Etanercept (Enbrel (Registered)) In Patients With Moderately Active Rheumatoid Arthritis In Every Day Clinical Practice In Austria
Brief Title: Study to Observe the Safety and Efficacy of Etanercept (Enbrel®) in Patients With Moderately Active Rheumatoid Arthritis in Every Day Clinical Practice in Austria
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801357
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Full Analysis Set: Full Analysis Set (FAS): The FAS contains any patient that has given written informed consent.
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — observation of Etanercept treatment in moderately active RA patients in Austria. Etanercept treatment according to Austrian SmPC

SUMMARY:
This is a prospective non-interventional observational study to evaluate the treatment of moderately active RA patients in every day clinical practice in Austria. Patients will be observed over 52 weeks. The primary endpoint will be percentage of patients who reach CDAI remission after 24 weeks.

DETAILED DESCRIPTION:
Non-interventional observational study, national, multicenter prospective non-interventional study (NIS) as defined by the Austrian Drug Law § 2a Section 3 N/A

ELIGIBILITY:
Inclusion Criteria:

1. The patient is eligible to receive Etanercept treatment according to the Austrian SmPC.
2. The decision to treat the patient with Etanercept has been made independently by the physician and is clearly separated from the decision to include the patient in the study. The treatment decision was made in advance and is not dependent on the protocol.
3. The patient was informed about the study and gave his/her consent and signed an Independent Ethics Committee (IEC) submitted written Informed Consent form on use of the data.
4. The patient has moderately active RA, defined as a disease activity of CDAI >10 and ≤22 and/or DAS28 (CRP)>3.2 and ≤ 5.1

Exclusion Criteria:

1. Any contraindication according to the Austrian SmPC, which includes:

   A hypersensitivity to any component of Etanercept, active tuberculosis or any other serious infection.
2. Patient has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderately active RA that are treated with Etanercept will be studied. All patients enrolled should meet the usual prescribing criteria for Etanercept as per the Austrian SmPC and should be entered into the study at the investigator's discretion.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2016-01-07 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Austria (10):
  - Ordination Dr. Thomas Muller, Graz
  - Barmherzige Brüder Graz Eggenberg, Graz
  - Ordination Dr. Horst Just, Klagenfurt
  - Ordination Dr. Richard Janetschko, Linz
  - Ordination Dr. Wilhelm Kaiser, Linz
  - Dr. Eichbauer-Sturm, Linz
  - Rheumazentrum Oberlaa, Vienna
  - Ordination Dr. Peter Peichl, Vienna
  - Ordination Dr. Maya Thun, Vienna
  - Ordination Dr. Thomas Schwingenschlogl, Wiener Neudorf

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801357&StudyName=Study%20to%20Observe%20the%20Safety%20and%20Efficacy%20of%20Etanercept%20%28enbrel%AE%29%20in%20Patients%20with%20Moderately%20Active%20Rheumatoid%20Arthritis%20in%20Every%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 111 participants were enrolled in the study but due to the loss of all study data and material at one site with 35 participants, the number of participants that could be included in the analysis was 76.
Groups:
- Etanercept: Participants with moderately active rheumatoid arthritis (RA), who received etanercept as per physician's discretion based on Austrian summary of product characteristics (SmPC) were observed prospectively up to Week 52. According to Austrian SmPC, recommended dose included etanercept 25 milligrams (mg) twice weekly, or 50 mg once weekly subcutaneous injection.
Period: Overall Study
Arm/Group | Etanercept
Started | 111
Treated | 76
Completed | 61
Not Completed | 50
Not completed — Adverse Event | 4
Not completed — Disease Remission | 1
Not completed — Withdrawal by Subject | 4
Not completed — Other | 2
Not completed — Lack of Efficacy | 4
Not completed — Data not available | 35

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included any participants who had given written informed consent.
Arm/Group | Etanercept
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Remission at Week 24
Description: CDAI is a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment), PtGA and PGA (assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0-76. CDAI less than equal to (<=) 2.8 indicates disease remission, greater than (>) 2.8 to 10 = low disease activity, greater than (>) 10 to 22 = moderate disease activity, and >22 = high disease activity. Percentage of participants with CDAI remission (score <=2.8) at Week 24 were reported.
Time Frame: Week 24
Population: Eligible Set included all participants who had given written informed consent and had received at least one dose of etanercept with evaluable CDAI assessments at baseline and Week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 61
percentage of participants | 44.3 [31.53 to 57.56]

2. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Status of Disease Activity at Week 12 and Week 52
Description: CDAI is a simplified index for assessing the disease activity comprising of the SJC, TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC, TJC (based on 28-joint assessment), PtGA and PGA (assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Percentage of participants with different type of CDAI status of disease activity (remission, low disease, moderate and high disease activity) at Week 12 and 52 were reported. Only those categories in which at least 1 participant had data were reported.
Time Frame: Week 12 and Week 52
Population: FAS included any participants who had given written informed consent.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 76
percentage of participants
  Remission At Week 12 | 22.4
  Low disease activity At Week 12 | 50.0
  Moderate disease activity At Week 12 | 11.8
  High disease activity At Week 12 | 2.6
  Remission At Week 52 | 48.7
  Low disease activity At Week 52 | 19.7
  Moderate disease activity At Week 52 | 7.9

3. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Scores at Week 12, Week 24 and Week 52
Description: CDAI is a simplified index for assessing the disease activity comprising of the SJC, TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC, TJC (based on 28-joint assessment), PtGA and PGA (assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: FAS included any participants who had given written informed consent. Here, "number analyzed" signifies participants who were evaluable at specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 76
units on a scale
  Baseline: number analyzed (Participants) | 71
  Baseline | 25.75 (8.195)
  Change at Week 12: number analyzed (Participants) | 61
  Change at Week 12 | -19.09 (7.903)
  Change at Week 24: number analyzed (Participants) | 61
  Change at Week 24 | -20.45 (8.746)
  Change at Week 52: number analyzed (Participants) | 55
  Change at Week 52 | -22.58 (7.732)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 8/76
Other Adverse Events (participants affected / at risk) | 16/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=76)
Atrial fibrillation (Cardiac disorders) | 2
Disease recurrence (General disorders) | 1
Borrelia infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=76)
Atrial fibrillation (Cardiac disorders) | 2
Disease recurrence (General disorders) | 1
Drug ineffective (General disorders) | 4
Injection site erythema (General disorders) | 1
Injection site rash (General disorders) | 1
Injection site reaction (General disorders) | 1
Borrelia infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.